CLINICAL TRIAL: NCT00004110
Title: Monoclonal Antibody 3F8 and Oral Etoposide for the Treatment of Neuroblastoma
Brief Title: Monoclonal Antibody Therapy Plus Etoposide in Treating Patients With Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: MSKCC-IRB-99033; CDR0000067333 (Registry Identifier: PDQ (Physician Data Query)); NCI-G99-1599
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Neuroblastoma
Keywords: regional neuroblastoma; disseminated neuroblastoma; recurrent neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — humanized 3F8 anti-GD2 monoclonal antibody; Etoposide; Isotretinoin

INTERVENTIONS:
Biological: monoclonal antibody 3F8
Drug: etoposide
Drug: isotretinoin

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody therapy plus etoposide in treating patients who have neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor effects of monoclonal antibody 3F8, etoposide, and isotretinoin using standard imaging methods and tumor marker studies in patients with high-risk neuroblastoma.
* Assess progression-free survival in these patients after this treatment.
* Assess the effects of oral etoposide on human anti-mouse antibody and anti-idiotype response in these patients.

OUTLINE: Patients are stratified according to disease status (evaluable but not measurable vs second or subsequent remission with no measurable or evaluable disease).

Patients receive monoclonal antibody 3F8 (MOAB 3F8) IV over 1.5 hours once daily on days 1-10 and oral etoposide once daily on days 29-49. Treatment repeats every 8 weeks for 4 courses in the absence of disease progression, human anti-mouse antibody (HAMA) response, or unacceptable toxicity.

If HAMA fails to develop after completion of 4 courses of MOAB 3F8, patients continue treatment with MOAB 3F8 on days 1-5 every 8 weeks until HAMA reaches greater than 1,000 U/mL or until month 24, whichever occurs first.

Beginning after completion of 4 courses of etoposide and MOAB 3F8 or if HAMA develops, patients receive oral isotretinoin twice daily for 14 days followed by at least a 14-day rest. Treatment repeats for a total of 6 courses.

PROJECTED ACCRUAL: A total of 50 patients (25 per stratum) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* High-risk neuroblastoma by:

  * Histopathology OR
  * Bone marrow involvement plus elevated urinary catecholamines
* Prior tumor progression on standard chemotherapy and poor long-term prognosis as indicated by 1 or more of the following:

  * N-myc amplification in tumor cells
  * Diploid chromosomal content plus lp loss of heterozygosity in tumor cells
  * Distant skeletal metastases
  * Unresectable primary tumor infiltrating across the midline
  * More than 10% tumor cells in bone marrow
  * Less than 30% chance of long-term progression-free survival
* Evaluable (microscopic marrow metastasis, elevated tumor markers, abnormal bone scan or MIBG or PET scan) but not measurable (CT scan, MRI) disease documented at least 4 weeks after completion of prior systemic therapy
* No rapidly progressive disease as defined by 1 or more of the following:

  * Serum lactic dehydrogenase greater than 1.5 times upper limit of normal due to tumor
  * An opiate requirement for pain from tumor
  * Greater than 25% increase in tumor by successive imaging studies
  * Life expectancy less than 8 weeks
* Second or subsequent remission after chemotherapy and/or radiotherapy allowed provided there is less than 30% chance of survival
* No prior myelodysplastic syndromes or leukemia

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* See Disease Characteristics
* At least 8 weeks

Hematopoietic:

* Not specified

Hepatic:

* No grade 3 or worse liver toxicity

Renal:

* No grade 3 or worse renal toxicity
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No grade 3 or worse cardiac toxicity

Pulmonary:

* No grade 3 or worse pulmonary toxicity

Other:

* Not pregnant
* No grade 3 or worse gastrointestinal toxicity
* No grade 3 or worse neurologic system toxicity
* No grade 4 hearing deficit
* No active life-threatening infection
* No prior exposure to mouse antibodies and human anti-mouse antibody greater than 1,000 ELISA units/mL
* No allergy to mouse proteins

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Kong V. Cheung, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States